CLINICAL TRIAL: NCT01062581
Title: University of Minnesota Transplant Registry
Status: Recruiting | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 0704M05324
Record Dates: First submitted 2010-02-03; First posted 2010-02-04 (Estimated); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Transplant Recipient; Transplant Donation
Keywords: Recipient; Donor; Organ Transplant; Registry; University of Minnesota

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Transplant Recipients and Living Donors: All transplant recipients receiving transplants at the University of Minnesota (kidney, pancreas, liver, heart, lung, islet, intestine). All ages.
  All living donors donating an organ at the University of Minnesota (kidney, pancreas, liver, lung) (by law, living donors are required to be at least 18 years old)

SUMMARY:
Under Transplant Information Services (TIS), the University of Minnesota Transplant Registry (UMTR) will serve as the repository for core research data.

DETAILED DESCRIPTION:
UMTR is a system of ongoing registration of cases seen in the transplant program at the University of Minnesota. The registry will: (1) provide core outcomes data and background information necessary to conduct outcomes management research in solid organ transplantation and advanced lung disease, and (2) support cutting edge research through existing program specific databases in liver, intestine, pancreas, islet, kidney, heart and lung transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Received a transplanted organ at the University of Minnesota
* Living donor who donates an organ at the University of Minnesota

Exclusion Criteria:

* Did not receive a transplant at the University of Minnesota
* Did not donate an organ at the University of Minnesota

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: University of Minnesota Transplant Center University of Minnesota Medical Center, Fairview
Sampling Method: Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 1997-03; Primary Completion 2050-01 (Estimated); Study Completion 2050-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Arthur Matas, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota Transplant Information Services, Minneapolis, Minnesota, United States